CLINICAL TRIAL: NCT05391256
Title: Referral of Callers to Retrieve Drone-delivered AEDs in Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Everdrone AB (Unknown); SOS Alarm AB (Unknown); Västra Götalandsregionen (Other); Green Flyway (Unknown); Aviation capacity resources AB (ACR) (Unknown); Region Jämtland Härjedalen (Other)
Responsible Party: Principal Investigator, Andreas Claesson, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRILL4
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Drone; AED; EMS; OHCA; UAV; Dispatch centre
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Automated flying Drone carrying an Automated external defibrillator (AED) (Experimental): Totally six drone systems are setup to be deployed in suspected OHCA cases as a complement to EMS. This is a single-arm intervention evaluating referral of bystanders during 112-calls to retrieve drone delivered AEDs in suspected OHCA.
  Interventions: Device: Automated flying Drone carrying an Automated external defibrillator (AED)

INTERVENTIONS:
Device: Automated flying Drone carrying an Automated external defibrillator (AED) — Totally n=6 drones are equipped with automated external defibrillators (AEDs). These drones are deployed by the dispatch centre to cases of suspected out-of-hospital cardiac (OHCA) as a complement to standard care (ambulance/EMS) over up to 12 months Monday to Sunday 08:00-22:00. The bystander onsite receives instructions from the dispatcher to retrieve the AED outside the house when it has been delivered by the drone. The bystander attaches the AED to the patients chest to facilitate early defibrillation.
  An interventional package directed to the dispatchers is distributed and consists of an e-learning program, an AED -trainer placed at the dispatch center. Within the dispatcher decision tool - there is information how to inform the caller to retrieve the AED. The HEMS-coordinator reminds the dispatcher during the call on operational information. Monthly information to staff of project progress is provided.

SUMMARY:
Time to defibrillation is the most important predictor of survival in cardiac arrest. Recent studies have shown that unmanned drones can deliver AEDs to the site of real life out-of hospital cardiac arrest (OHCA) before ambulance arrival. Although an AED is available in the close vicinity, they are seldom used. The overall aim of this study is to provide an interventional bundle directed towards the dispatch centre and evaluate referral of callers to retrieve drone-delivered AEDs so that they may be attached in cases out-of-hospital cardiac arrest.

DETAILED DESCRIPTION:
This is an observational, non-randomized single group assignment study with the primary purpose of evaluating Referral of callers to retrieve drone-delivered AEDs in out-of-hospital cardiac arrest.

Totally, six AED-equipped drones will be placed in hangars at six different sites covering a geographic area of about 230 km2 and approximately 150,000 inhabitants for dispatch to suspected cases of OHCA as a complement to standard care i.e., ambulance. By coordinating the operations with local Air Traffic Control (ATC), the risk of airspace conflicts, or in worst case collisions, is mitigated to an acceptable level.

The investigators estimate to enroll some 150 alerts and 60 participants during a study period of up to 12 months. The investigators will closely follow and study the potential of dispatcher referral of 112-callers to retrieve and use drone delivered AEDs prior ambulance arrival.

The drone operator, Everdrone, has integrated all software and hardware for the concept on the DJI Matrice 600 Pro drone. Examples of added features: an integrated Parachute Rescue System (validated by independent third party using the ASTM F3322 - 18 standard), a high precision sense and avoid system and a winching device to safely lower the AED to ground at delivery from 30 meters altitude. Furthermore, Everdrone AB has fully integrated their system and operational routines with the dispatch central, emergency medical services and aviation organizations. As a result from previous study (version 1.0) a number of hardware and software improvements have been made to the system (version 2.0).

Six hangars are setup at optimal locations in each of the six administrative areas. Hangars are large isolated tents 4x4 meters in where the drone is placed, remotely operated and surveiled by camera. Hangars are within fenced areas so that the public has no access. They are equipped with weather stations and an automated gate which automatically will open on alert.

When an emergency 112-call is answered it is indexed by the dispatcher depending on the patients condition. If an OHCA is suspected, the dispatcher indexes the event as a)"ongoing cardio-pulmonary resuscitation (CPR)" or b) "Unconscious with abnormal or absent breathing". If an emergency call is identified within administrative areas AND indexed as "a" or "b" an automated (not manual as with ambulance alerts) alert is sent via radio-alert to the drone operator. This triggers:

boot-up of the drone drone hangar gate opening route-planning of the mission weather condition confirmation remote pilot acceptance of the mission remote pilot calling ATC for takeoff approval

The drone system receives an alert from the dispatch center and the drone takes off from the hangar after approval from the drone pilot. For safety reasons all beyond visual line of sight (BVLOS) flights are done within the controlled airspace of Säve airport, Malöga airport and Östersund airport. Approval from ATC is granted for every single flight. Each flight will be carried out at 60-80 meters of altitude, have a preliminary maximum flight speed of 70 km/h, and a maximum range of 6 km one-way. The drone system is remotely deployed and surveiled from the drone operating center at Everdrone. The drone is dispatched alongside ambulance as a complement to standard care. The drone systems are designed to operate in dry conditions with median winds not exceeding 8 m/s and during both day and night conditions.

The AED used is an ultra-light AED (FRED Easyport from Schiller), weighting totally 800 grams with basket and siren. Upon arrival onsite the basket with the AED will be winched down from about 30 m altitude and delivered within 10 meters from the object i.e., the front door or onsite in public areas. Local AED drone support after completed mission includes electrode change battery test, potentially pic-up up the drone after dispatch by the Everdrone personnel.

Dispatch of the drone in suspected OHCA cases will be executed as a complement to standard care i.e., ambulance between 1 June 2022 to 31 May 2023, totally up to 12 months of full-scale real-life flights to suspected OHCA victims. Based on historical data of OHCA from the Swedish register for cardiopulmonary resuscitation (SRCR) and first ever dispatch of AED-equipped drones during 2020 the drone systems will be alerted in an estimated 150 cases (about 3 flights/ week) of suspected OHCA over the study period. Predefined exclusion criteria (rain, median wind > 8 m/s, high rise buildings >20m, pre-flight checklists not OK) will presumably prohibit flights, thus making an estimated 60 cases eligible for inclusion (i.e., drone takes off and delivers an AEDs in suspected OHCA.)

All cases where an AED is delivered by a drone prior to EMS arrival will be included in the study. An interventional package directed to the dispatchers is distributed from May 2022 and onwards and consists of an e-learning program, an AED -trainer placed at the dispatch center. Within the dispatcher decision tool - there is information how to inform the caller to retrieve the AED. The HEMS-coordinator reminds the dispatcher during the call that the drone is on its way and after delivery of the AED and as well on operational information such as drop-spot. Monthly information to staff of project progress is provided.

The dispatcher will try to refer the caller to retrieve the drone-delivered AED, the bystander will be encouraged to physically collect/retrieve the AED so that it may be attached to the patient suffering from OHCA.

Dispatchers compliance to the routine of referring callers to retrieve the drone-delivered AED so that it may be attached to the patient is evaluated from start of the project June 2020 to May 2023. Interventions directed towards the dispatch center will be described in chronological order in relation to the outcome parameters proportion (percentages) of referral, retrieval and attachment of AEDs.

ELIGIBILITY:
Inclusion Criteria:

* All suspected OHCA during 112-calls including drowning
* Within prespecified administrative areas (excluding no delivery- and no-fly zones)
* Hours of operation: 08:00-22:00 (daylight conditions)
* Drone system online

Exclusion Criteria:

Pre-alert:

* Children <8 years
* Trauma
* EMS-witnessed cases

Post alert:

* ATC non-approval of flight
* Rain, winds exceeding 8m/s (median)

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion (percent) of cases where a bystander attaches a drone-delivered AED to the OHCA- patients chest, prior the arrival of EMS. | Up to 12 months
  In all alerts to suspected OHCA where a drone took off and delivered an AED on the ground, all cases were a bystander attaches the drone delivered AED to the OHCA-patients chest as instructed in T-CPR protocol before ambulance arrival will be measured. In all alerts to suspected OHCA where a drone took off and delivered an AED on the ground, all cases were a bystander attaches the drone delivered AED to the OHCA-patients chest as instructed in T-CPR protocol before ambulance arrival will be measured. Percentages.

SECONDARY OUTCOMES:
Proportion (percent) of cases where a dispatcher verbally refers a bystander to retrieve a drone-delivered AED on the ground before EMS arrival in cases of OHCA | Up to 12 months
  In all alerts to suspected OHCA where a drone took off and delivered an AED on the ground, the dispatcher verbally tries to refer the bystander to retrieve the drone delivered AED before ambulance arrival. Proportion of cases where the dispatcher tries to refer the caller is measures (percentages). Accurate completion of mission is defined as delivery of an AED onsite on the ground in close connection from the OHCA, AEDs is accessible to the bystander and the dispatcher refers the caller to retrieve the AED through T-CPR instructions.
Proportion (percent) of cases where a bystander successfully retrieves a drone-delivered AED from the ground as instructed by the dispatcher. | Up to 12 months
  In all alerts to suspected OHCA where a drone took off and delivered an AED on the ground, the bystander physically retrieves the drone-delivered AED as instructed by the dispatcher during T-CPR before ambulance arrival. All cases with successful retrieval of the AED will be measured (percentages).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Claesson, Ph.D, Principal Investigator — Department of Clinical Science and Education, Södersjukhuset, Karolinska institutet
Locations (2):
- Sweden (2):
  - Region Jämtland, Östersund, Jämtland County
  - Västra Götalandsregionen, Gothenburg, VGRegion

IPD SHARING:
Plan to Share IPD: No